CLINICAL TRIAL: NCT00439959
Title: A Double-Blind, Parallel, Randomized, Placebo-Controlled, Single and Repeat Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK625433 in Healthy Subjects and in Subjects Who Are Chronically Infected With Hepatitis C.
Brief Title: Monotherapy Versus Placebo Over 14 or 17 Days in Healthy and Hepatitis C Infected Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: HSP108233
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-03

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
Keywords: GSK625433,; Hepatitis C,; metabolic probe,; food-effect,; HCV,; FTIH; polymerase,
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK625433/placebo

SUMMARY:
This study represents the first administration of GSK625433 in humans. The study is designed to evaluate initial safety and tolerability in healthy adults as well as anti-viral activity in Hepatitis C(HVC) infected adults. The way the human body processes GSK625433 will also be investigated.

ELIGIBILITY:
Inclusion criteria:

* Healthy males & females
* Part 1 ages 18-60
* Part 2 ages 18-50 & 65-80
* Within normal weight range given your height
* Negative urine drug and alcohol test
* Willing to follow all study procedures

Exclusion criteria:

* Any significant abnormal lab, ECG, medical or physical exam finding during screening
* Allergy to the study drug
* Excessive alcohol intake
* Positive HIV or hepatitis B or C result
* Use of prescription or non-prescription drugs within one week of study start except for birth control
* Blood pressure meds & Tylenol
* Pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-10; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Safety parameters: adverse events; telemetry; clinical laboratory values, vital signs, and ECGs. Plasma levels of GSK625433. Change in HCV viral load. Taken throughout the study | 17 Days

SECONDARY OUTCOMES:
Plasma levels of GSK625433. Metabolic analysis of CYP substrates to estimate enzyme activity. Resistance analysis for subjects with HCV infection. Taken throughout the study | 17 Days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Evansville, Indiana, United States